CLINICAL TRIAL: NCT06276127
Title: Oral Bisoprolol Versus Intravenous Diltiazem in the Management of Atrial Fibrillation or Flutter With Rapid Ventricular Rate in the Emergency Department: A Randomized Controlled Trial
Brief Title: Oral Bisoprolol Vs IV Diltiazem in Atrial Fibrillation or Flutter With Rapid Ventricular Rate.
Acronym: BisoAF
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Fatin Khalfan Alomairi, Resident, Emergency Medicine, OMSB, Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MERC301123
Record Dates: First submitted 2024-02-18; First posted 2024-02-23 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation With Rapid Ventricular Response; Atrial Flutter With Rapid Ventricular Response
Keywords: Bisoprolol; AF; Diltiazem; Atrial flutter
MeSH Terms: conditions — Atrial Flutter | interventions — Bisoprolol

STUDY DESIGN:
Intervention Model Description: Study Design: Open-label, randomized controlled trial.
  Participants: Patients with atrial fibrillation/flutter and rapid ventricular rate.
  Treatment Arms: Oral Bisoprolol vs. Intravenous Diltiazem.
  Randomization: Subjects randomly assigned to either treatment group.
  Primary Endpoint: Reduction of heart rate to a target level within a specific timeframe.
  Secondary Outcomes: Adverse effects, hospital admission rates, additional rate control needs.
  Objective: Compare effectiveness and safety of oral Bisoprolol to intravenous Diltiazem.
  Monitoring: Continuous observation of vital signs and electrocardiograms for safety.
Masking Description: While the treating physician, nurse, and the patient will not be blinded to the treatment, the statistician analyzing it will remain blinded to treatment allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Bisoprolol (Experimental): A single oral dose of 5 mg Bisoprolol (maximum dose of 5 mg)
  Interventions: Drug: Oral Bisoprolol
- Intravenous Diltiazem (Other): single intravenous dose of Diltiazem at 0.25 mg/kg (to a maximum dose of 30 mg)
  Interventions: Drug: Intravenous Diltiazem

INTERVENTIONS:
Drug: Oral Bisoprolol — Participants in this group will receive a single oral dose of Bisoprolol, set at a dosage of 5 mg, with a maximum dose limit of 5 mg.
  Other Names: Bisoprolol hemifumarate
  Arms: Oral Bisoprolol
Drug: Intravenous Diltiazem — Participants in this group will be administered a single intravenous dose of diltiazem at a dosage of 0.25 mg/kg, with a maximum dose capped at 30 mg.
  Other Names: Diltiazem nondihydropyridine calcium channel blocker
  Arms: Intravenous Diltiazem

SUMMARY:
INTRODUCTION: The study focuses on comparing the effectiveness of oral Bisoprolol, a beta-1 adrenergic receptor blocker, against intravenous Diltiazem, a calcium channel blocker, in treating rapid atrial fibrillation or flutter with rapid ventricular response in an emergency setting. This research aims to fill the gap in empirical evidence regarding the use of oral Bisoprolol for these conditions, potentially offering a convenient, evidence-based alternative for patient management in emergency departments where established protocols are lacking.

METHOD: This study is a randomized controlled trial targeting patients who present to the emergency room with symptomatic atrial fibrillation or flutter and rapid ventricular response requiring intervention. Participants will be split into two groups and undergo continuous monitoring of vital signs and regular electrocardiograms to ensure safety and document any adverse effects. The primary focus is on patient safety while evaluating the efficacy of the treatments.

AIM: Evaluate the efficacy and safety of oral bisoprolol in treating atrial fibrillation or atrial flutter with rapid ventricular response in an emergency department setting.

PRIMARY OJECTIVES: The primary efficacy outcome will be evaluated by achieving a HR<110 beats per minute or a decrease ≥20% of baseline HR at 60 minutes. The primary safety outcome measures are HR < 60 bpm and SBP < 95 mm Hg.

SECONDARY OBJECTIVES: The use of Rescue medication, proportion of patients who required hospitalization, worsening of heart failure or pulmonary oedema, side effect of medication ( dizziness, headaches, gastrointestinal symptoms)

PATEINT POPULATION: Adults (18 and older) presenting to the emergency department at Sultan Qaboos University Hospital with symptomatic atrial fibrillation or atrial flutter with rapid ventricular response requiring treatment.

INTERVENTION: A single oral dose of 5 mg Bisoprolol (maximum dose of 5 mg) or a single intravenous dose of Diltiazem at 0.25 mg/kg (to a maximum dose of 30 mg).

CLINICAL MEASURMENT: Heart rate recorded every 15 minutes up to the 90-minute mark, with a 12-lead ECG performed every 30 minutes.

OUTCOME: For therapy to be considered effective, patients must achieve a ventricular rate ≤110/min or experience a drop-in ventricular rate of at least 20% at 60 minutes.

DETAILED DESCRIPTION:
= Aim of the Study: This open-label randomized controlled trial (RCT) aims to assess the effectiveness and safety of oral bisoprolol in treating atrial fibrillation (AF) with rapid ventricular response (RVR) and atrial flutter within an acute ED setting. We aim to determine the viability of utilizing oral bisoprolol as a primary treatment option for atrial fibrillation with rapid ventricular response (RVR) and atrial flutter by evaluating its clinical outcomes, focusing on rate control and potential adverse effects, and comparing them with those of intravenous diltiazem. The findings from this research will enhance our understanding and guide clinicians towards evidence-based therapeutic decisions, ensuring optimal patient care and improved outcomes.

= Research Objectives and Hypothesis: The research aims to test the null hypothesis, which posits that there is no significant difference in achieving a heart rate (HR) below 110 beats/min or a reduction in ventricular rate by at least 20% between the oral bisoprolol (PO) and intravenous diltiazem (IV) groups after 60 minutes.

= Study Design: This is a prospective, open-label, randomized controlled trial that will be conducted as a single-center investigation within the Emergency Department of Sultan Qaboos University Hospital (SQUH). This study will involve adult patients aged 18 and older, and all eligible participants will be given written informed consent to join the research.

= Control Group: Participants in this group will be administered a single intravenous dose of diltiazem at a dosage of 0.25 mg/kg, with a maximum dose capped at 30 mg.

= Intervention Group: Participants in this group will receive a single oral dose of bisoprolol, set at a dosage of 5 mg, with a maximum dose limit of 5 mg.

* Primary Endpoints:

  * The primary efficacy outcome evaluated by achieving a HR < 110 beats per minute or a decrease ≥20% of baseline HR at 60 minutes.
  * The primary safety outcome measures were HR < 60 bpm and SBP < 95 mm Hg.
* Secondary Endpoints:

  * The use of rescue medication (Rescue rate control defined as the administration of a supplementary rate control medication after 60 minutes of the initial dose of the interventional drug).
  * Proportion of patients who required hospitalization (hospital admission/ICU admission).
  * ED revisit.
  * Treatment-related adverse events.
  * Dizziness, headaches, gastrointestinal symptoms.
  * Worsening of heart failure or pulmonary edema.
* Sample Size:

In addressing the novel concept of comparing the effectiveness of oral bisoprolol versus IV diltiazem in treating AF or atrial flutter with RVR in an acute setting, we aim to conduct a pilot study with 30 patients in each group to calculate the study sample size.

* Study Procedures:

  1. Present to the Clinical Site:

     * An eligible adult patient aged 18 years or older, who presents with symptomatic rapid ventricular response atrial fibrillation or atrial flutter and requires treatment for rate control.
  2. Eligibility Assessments:

     * Inclusion and exclusion criteria will be checked.
  3. Informed Consent:

     * Potentially eligible participants will be identified by their treating clinicians. Written informed consent to participate in this study will follow a process of information exchange between clinicians and potential participants.
  4. Study the Effectiveness in Achieving Rate Control:

     * Data will be collected prospectively, including demographics, medical history, vital signs, and ECG results. Each patient will be promptly assessed, and continuous monitoring will be established for every patient to monitor cardiac rhythm, heart rate (HR), blood pressure, and oxygen saturation levels.
     * Heart rate will be recorded every 15 mins till the 90-minute mark.
     * For the therapy to be considered effective, the patients had to achieve a ventricular rate ≤110/min or experience a drop in ventricular rate of at least 20% at 60 minutes.
     * 12-lead ECG will be done every 30 minutes at 0, 30, and 60 minutes.
     * Relevant secondary outcomes will be recorded.
  5. Standard-of-Care Procedures:

     * Patients may receive additional medications as part of their emergency department treatment after 60 minutes if they remain hemodynamically stable. Any additional medications administered will be recorded. The need for additional medications (including the drug administered, the dose, the time, and the route of administration) will be recorded.
  6. Safety Assessments:

     * All adverse events will be documented on the adverse event case log. Serious adverse events should be immediately reported to the primary investigator. Any serious adverse event will be reported immediately to the Institutional Review Board. An adverse event is considered serious if it causes a threat to the patient's life or functioning. The U.S. Food and Drug Administration (FDA) defines a serious adverse event (SAE) as any untoward medical occurrence that:
     * Results in death.
     * Is life-threatening (places the patient at risk of death).
     * Requires hospitalization or prolongs an existing hospitalization.
     * Causes persistent or significant disability or incapacity.
     * Requires medical intervention to prevent one of the above outcomes.
  7. Follow-Up:

     * All participants will be followed up after 24 hours and 48 hours.
* Risks and Benefits:

Bisoprolol, a cardioselective beta-1 adrenergic agent, is recognized for its potency and the convenience of once-daily dosing. It is well-tolerated and deemed suitable for patients with chronic bronchoconstrictive disease, with safety established through clinical trials. On the other hand, diltiazem, a calcium channel blocker, is commonly used for hypertension and short-term AF management due to its rapid onset and lower impact on blood pressure, making it suitable for emergencies.

In collaboration with cardiology experts, the designated 60-minute time frame has been established to balance clinical relevance with patient safety. The administration of oral bisoprolol is considered a reliable and convenient treatment modality, assumed to be fast, painless, and associated with a lower risk of complications. This approach aims to facilitate a smooth transition to oral maintenance and provide an alternative for AF management in a busy Emergency Department. Meanwhile, intravenous (IV) diltiazem is acknowledged for its rapid onset, rendering it effective for the treatment of symptomatic atrial fibrillation patients in the emergency department. Throughout the ED phase, each patient will undergo close monitoring to ensure their utmost safety.

It is crucial to carefully consider the balance between potential benefits and risks, particularly in cases involving heart failure patients. Detailed monitoring protocols are in place to swiftly detect and manage any adverse effects or complications that may arise. Our preemptive strategies include comprehensive and regular patient monitoring, the implementation of an emergency protocol to address unexpected issues, and a meticulous medication review prior to any treatment administration. We are committed to transparent and ongoing communication with all study participants, maintaining a continuous focus on safeguarding their health and ensuring that the potential advantages of participation outweigh the risks.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old.
* Atrial fibrillation (RVR) or Atrial flutter on electrocardiogram.
* Heart rate >120 beats/min
* Stable patient with stable vital signs (Defined as having a SBP >110 mmHg, oxygen saturation > 94% on room air or with a simple face mask, a respiratory rate within normal limits, being conscious and oriented, and not having any concurrent life-threatening conditions such as myocardial infarction (MI) or Class IV heart failure).
* Mentally competent patient who can understand and sign the consent form.

Exclusion Criteria:

* Acute myocardial infarction.
* Known congenital and acquired valvular defects.
* Pre-excitation syndromes.
* Ventricular rate > 220beats/min.
* Administration of AV nodal blocking agents within the previous 24 h (beta blockers, non-dihydropyridine calcium channel blockers, digoxin and amiodarone or receiving regular maintains oral dose).
* Allergy to either bisoprolol or diltiazem.
* Severe hepatic and renal failure.
* Pregnancy / breastfeeding.
* A history of cocaine or methamphetamine use within 24 hours before arrival.
* Known Asthmatic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy Outcome Evaluated by Achieving the Target Heart Rate Reduction | at 60 minutes
  The primary efficacy outcome evaluated by achieving a HR<110 beats per minute or a decrease ≥20% of baseline HR at 60 minutes
Safety Outcome Evaluated by the Presence of serious adverse event | at 60 minutes
  The primary safety outcome measures were HR < 60 bpm and SBP < 95 mm Hg

SECONDARY OUTCOMES:
The use of Rescue medication | 60 minutes
  Rescue rate control defined as the administration of a supplementary rate control medication after 60 minutes of the initial dose of the interventional drug
Proportion of patients who required hospitalization | 90 minutes
  percentage of individuals within a study who need to be admitted to a hospital for treatment, observation, or further medical care
ED revisit | First 48 hour from discharge
  Number of patient who will revisit ED with symptomatic AF after stabilization and discharge
Number of Participants Experiencing Treatment-Related Adverse Events | First 48 hour after receive intervention
  Any patient experience ( Dizziness, headaches, gastrointestinal symptoms , Worsening of heart failure or pulmonary edema )

CONTACTS AND LOCATIONS:
Overall Officials: Usama Al Khalasi, MD, Study Chair — The Medical City for Military & Security Services, Oman
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Al-khod, Oman

IPD SHARING:
Plan to Share IPD: Yes
Will share the Study Protocol and Statistical Analysis Plan (SAP) to enhance transparency and provide detailed insights into our study's design, methodologies, statistical analyses, and inclusion criteria.
Supporting Information: Study Protocol, SAP
Time Frame: Data from our study will be available soon after its completion and will remain accessible for a period of 3 years.
Access Criteria: Open Access Policy: The document is accessible to anyone who requests it, promoting widespread dissemination.

REFERENCES:
- [Background] Fromm C, Suau SJ, Cohen V, Likourezos A, Jellinek-Cohen S, Rose J, Marshall J. Diltiazem vs. Metoprolol in the Management of Atrial Fibrillation or Flutter with Rapid Ventricular Rate in the Emergency Department. J Emerg Med. 2015 Aug;49(2):175-82. doi: 10.1016/j.jemermed.2015.01.014. Epub 2015 Apr 22. PMID 25913166
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Posen A, Bursua A, Petzel R. DOsing Strategy Effectiveness of Diltiazem in Atrial Fibrillation With Rapid Ventricular Response. Ann Emerg Med. 2023 Mar;81(3):288-296. doi: 10.1016/j.annemergmed.2022.08.462. Epub 2022 Nov 17. PMID 36402632
- [Background] Saksena S, Slee A, Waldo AL, Freemantle N, Reynolds M, Rosenberg Y, Rathod S, Grant S, Thomas E, Wyse DG. Cardiovascular outcomes in the AFFIRM Trial (Atrial Fibrillation Follow-Up Investigation of Rhythm Management). An assessment of individual antiarrhythmic drug therapies compared with rate control with propensity score-matched analyses. J Am Coll Cardiol. 2011 Nov 1;58(19):1975-85. doi: 10.1016/j.jacc.2011.07.036. PMID 22032709
- [Background] Groenveld HF, Crijns HJ, Tijssen JG, Alings M, Hillege HL, Tuininga YS, Van den Berg MP, Van Veldhuisen DJ, Van Gelder IC. Rate control in atrial fibrillation, insight into the RACE II study. Neth Heart J. 2013 Apr;21(4):199-204. doi: 10.1007/s12471-013-0391-1. No abstract available. PMID 23468405
- [Background] Bakheit AH, Ali R, Alshahrani AD, El-Azab AS. Bisoprolol: A comprehensive profile. Profiles Drug Subst Excip Relat Methodol. 2021;46:51-89. doi: 10.1016/bs.podrm.2020.07.006. Epub 2020 Sep 8. PMID 33461700
- [Background] clinical_evaluation_of_bisoprolol_in_the_treatment.31.
- [Background] Ishiguro H, Ikeda T, Abe A, Tsukada T, Mera H, Nakamura K, Yusu S, Yoshino H. Antiarrhythmic effect of bisoprolol, a highly selective beta1-blocker, in patients with paroxysmal atrial fibrillation. Int Heart J. 2008 May;49(3):281-93. doi: 10.1536/ihj.49.281. PMID 18612186
- [Background] A randomized trial of beta-blockade in heart failure. The Cardiac Insufficiency Bisoprolol Study (CIBIS). CIBIS Investigators and Committees. Circulation. 1994 Oct;90(4):1765-73. doi: 10.1161/01.cir.90.4.1765. PMID 7923660
- [Background] The Cardiac Insufficiency Bisoprolol Study II (CIBIS-II)-.
- [Background] Demircan C, Cikriklar HI, Engindeniz Z, Cebicci H, Atar N, Guler V, Unlu EO, Ozdemir B. Comparison of the effectiveness of intravenous diltiazem and metoprolol in the management of rapid ventricular rate in atrial fibrillation. Emerg Med J. 2005 Jun;22(6):411-4. doi: 10.1136/emj.2003.012047. PMID 15911947
- [Background] Hasbrouck M, Nguyen TT. Acute management of atrial fibrillation in congestive heart failure with reduced ejection fraction in the emergency department. Am J Emerg Med. 2022 Aug;58:39-42. doi: 10.1016/j.ajem.2022.03.058. Epub 2022 Apr 6. PMID 35623182
- [Background] Nicholson J, Czosnowski Q, Flack T, Pang PS, Billups K. Hemodynamic comparison of intravenous push diltiazem versus metoprolol for atrial fibrillation rate control. Am J Emerg Med. 2020 Sep;38(9):1879-1883. doi: 10.1016/j.ajem.2020.06.034. Epub 2020 Jun 21. PMID 32745920
- See also: Lawrence Rosenthal MPFFP of MDS of CP and ED of EFPD of CDU of MMMC. Atrial Flutter. — https://emedicine.medscape.com/article/151210-overview
- See also: Diltiazem — https://go.drugbank.com/drugs/DB00343